CLINICAL TRIAL: NCT05996939
Title: Effectiveness of Unstable Shoes on Volume and Quality of Life in Lower Limb Lymphedema.
Brief Title: Use of the Unstable Shoes in Lower Limb Lymphedema.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Vanesa Abuín, Doctor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UEM_LIN_2011_01
Record Dates: First submitted 2023-07-28; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Lower Limb Lymphedema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unstable shoes (Experimental): Use of unstable shoes for 8 weeks
  Interventions: Other: To compare the efficacy of unstable shoes with that of conventional sports shoes in people with lower-limb primary and secondary lymphedema.
- Usual sports footwear (No Intervention): Use of conventional shoes for 8 weeks

INTERVENTIONS:
Other: To compare the efficacy of unstable shoes with that of conventional sports shoes in people with lower-limb primary and secondary lymphedema. — Unstable shoes were compared with conventional sports shoes, the objective being to evaluate possible differences in the evolution of lymphedema. During a clinical trial lasting eight weeks, we assessed quality of life, limb volume, and symptoms derived from lymphedema.
  Arms: Unstable shoes

SUMMARY:
Lymphedema is an external manifestation of lymphatic system insufficiency and deranged lymph transport. It is defined as accumulation in the extracellular space of protein-rich fluid, due to a mechanical failure of the lymphatic system. Lymphedema directly affects the quality of life of the patient, not only in the physical aspect, but also in the psychological, sexual and social aspects. Muscle and joint pumps are important external mechanisms of lymphatic and venous fluid return improvement. The unstable shoes demands, especially during standing, increased muscle activity in the lower extremities. A clinical trial was carried out comparing both kinds of footwear, the objective being to evaluate possible differences in the evolution of lymphedema. Unstable shoes (MBT®) were compared with conventional sports shoes. During a clinical trial lasting eight weeks, we assessed quality of life, limb volume, and symptoms derived from lymphedema. The results suggested that the use of unstable shoes is recommendable for walking and for long periods of standing, since it decreases leg cramping and paraesthesia of affected limbs.

DETAILED DESCRIPTION:
Participants Subjects were recruited amongst the members of a Spanish association of people affected with lymphedema. Inclusion criteria were a) Subjects affected with lower limb lymphedema -primary, secondary, unilateral or bilateral-, b) Daily use of a compression stocking. Exclusion criteria were a) Subjects with acute infection of the affected limb b) that did not had any treatment for lymphedema one year prior to the study, c) Weight <40kg, d) shoe size <EU35 or >EU47 e)that have previously used unstable shoes f) vestibular alterations, vertigo, hypoacusis c) visual compromise that affects balance.

Procedure Written informed consent was obtained from the participants before the intervention. Random allocation to experimental and control group, was performed using Excel built-in function RAND ().. The generated sequence was employed to allocate the participants to one of the trial groups (e.g., intervention or control). Participants followed an 8 week intervention. Experimental group (EG) were provided with unstable sole shoes (MBT®, Masai Barefoot Technology Spain SL,08021 Spain.) and asked to wear them following a standardized protocol: 1 hour on day 1, increasing 1h each 2 days until 4h of daily use are achieved, during standing position and walking in the context of daily live activities, excluding sport activities. Control group (CG) was provided with a conventional sole sports footwear, following the same protocol that EG.

Outcome measures Circumferencial measure. Circumferencial measure was evaluated using a tape measure to measure the circumference of the foot at different points. Distal (4 cm from the base of the nail towards proximal) and Proximal (4 cm from the previous measurement).

Volume. Kuhnke's formula was used to calculate the estimated volume of the affected limb(241) V=(C12 + C22 +… Cn2)/π, Where V represents the volume and C refers to the different diameters of the limb, measured in centimeters.

Perception of the participants' clinical manifestations (243): measured through a questionnaire on perception of the state of the person's vascular alteration referred to the affected limb. In this survey, the subject is asked to value their symptoms (included heaviness, spider veins, swelling, pain, appearance of varicose veins, cramps, paresthesia and venous ulcers) with a 4-point scale: 0=absent, 1=mild/moderate, 2=important, 3=severe. In addition to lower limb swelling, other important symptoms experienced are heaviness, tightness, and pain. As there is no validated scale or survey to measure these symptoms characteristic of lymphedema, we used as a reference a previous study [10], where the symptoms or clinical manifestations compatible with chronic venous insufficiency that can be extrapolated to lymphedema are described.

In addition, a Change of habits survey was conducted at the end of the intervention period

ELIGIBILITY:
Inclusion Criteria:

-Subjects affected with lower limb lymphedema -primary, secondary, unilateral or bilateral-, -Daily use of a compression stocking

Exclusion Criteria:

* Subjects with acute infection of the affected limb
* that did not had any treatment for lymphedema one year prior to the study,
* Weight <40kg,
* shoe size <EU35 or >EU47
* that have previously used unstable shoes
* vestibular alterations, vertigo, hypoacusis
* visual compromise that affects balanc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Volume of the lower limb | 8 weeks
  Volume of the lower limb

SECONDARY OUTCOMES:
Circumference measure of the foot | 8 weeks
  Circumference measure of the foot
Changes in lymphedema symptoms | 8 weeks
  Changes in lymphedema symptoms